CLINICAL TRIAL: NCT03458117
Title: A Phase I, Open Label, Single Arm, Single Centre Study to Evaluate Mechanism of Action of Talimogene Laherparepvec (T-VEC) in Locally Advanced Non-melanoma Skin Cancer
Brief Title: T-VEC in Non-melanoma Skin Cancer
Acronym: 20139157 T-VEC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20139157
Record Dates: First submitted 2018-02-19; First posted 2018-03-08 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Non-melanoma Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma; Cutaneous Lymphoma; Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Lymphoma, T-Cell, Cutaneous; Carcinoma, Merkel Cell | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Talimogene Laherparepvec (T-VEC) (Experimental): Intralesional injections of T-VEC up to 4.0 mL of 10 to the 6 plaque-forming Units/mL (PFU/mL)
  Interventions: Genetic: Talimogene Laherparepvec (T-VEC)

INTERVENTIONS:
Genetic: Talimogene Laherparepvec (T-VEC) — a modified herpes simplex virus-1 (HSV-1) containing the gene coding for human granulocyte macrophage colony-stimulating factor (GM-CSF)

SUMMARY:
Evaluation of the mechanism of Action of talimogene laherparepvec (T-VEC) in patients with locally advanced non-melanoma skin cancer.

DETAILED DESCRIPTION:
This study evaluates the administration of T-VEC in non-melanoma skin cancer. The aim is to evaluate the effectiveness, safety and tolerability of T-VEC in patients with non-melanoma skin cancer through determination of local immune effects after repeated T-VEC injections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects Age ≥ 18 years
* histologically confirmed diagnosis of locally advanced squamous cell carcinoma, basal cell, carcinoma, Merkel cell carcinoma or cutaneous T cell lymphoma
* at least 1 injectable cutaneous lesion ≥ 20 mm in longest Diameter or multiple injectable lesions that in Aggregate have a longest Diameter of ≥ 50 mm
* Eastern Cooperative Oncology Group-Status (ECOG Status) 0 or 1
* Adequate organ functions

Exclusion Criteria:

* Hypersensitivity to T-VEC or any of ist components
* Presence of organ and lymph node metastases
* history or evidence of active autoimmune disease that requires systemic Treatment
* Evidence of clinically significant immunosuppression
* active herpetic skin lesions or prior complications hereof
* pregnancy, breast feeding
* requires intermittent or chronic systemic Treatment with an antiherpetic drug
* acute or chronic active Hepatitis B or C infection or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline local immune effects after repeated T-VEC injections | at baseline, after 3 injections (week 6) and optionally after 6 injections (week 12)
  Detection of increased local immune activation markers in skin biopsies of injected lesions. The following markers will be assessed by Polymerase chain reaction (PCR): interferon (IFN), 2-prime, 5-prime oligoadenylate synthetase 1 (OAS1), Interferon-induced GTP-binding protein MxA (MXA) and C-X-C motif chemokine 11 (CXCL11)

SECONDARY OUTCOMES:
Detection of Tumor Regression using World Health Organization (WHO) response criteria | at baseline and at week 22
  Measurement of the treated tumor size will be performed at baseline and at each visit until end of the study
Systemic immune response | at baseline and week 6, optionally also at week 12
  Detection of increased systemic immune Response markers in sera and peripheral blood mononuclear cells by multi-Color fluorescence-activated cell sorting (FACS)
Analysis of Adverse events | At week 1, 4, 6, 8, 10, 12, 14, 16, 18, 22
  All serious and non-serious adverse events that occur after enrollment through 30 (+7) days after the last administration of T-VEC will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, Prof. Dr., Principal Investigator — vice-director dermatology
Locations (1):
- Department of Dermatology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No